CLINICAL TRIAL: NCT05529290
Title: Evaluation of the Efficacy of Different Drugs in the Treatment of the Pain in Patients With Temporomandibular Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03.07.2019/10
Record Dates: First submitted 2022-02-14; First posted 2022-09-07 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — dexketoprofen trometamol; thiocolchicoside; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexketoprofen Trometamol + Thiocolchicoside (Active Comparator): (25mg + 4mg, 2x1)
  Interventions: Drug: Dexketoprofen Trometamol + Thiocolchicoside
- Dexketoprofen Trometamol + Paracetamol (Active Comparator): (25mg + 300mg, 2x1)
  Interventions: Drug: Dexketoprofen Trometamol + Paracetamol
- Dexketoprofen Trometamol (Active Comparator): (25mg, 2x1)
  Interventions: Drug: Dexketoprofen Trometamol (25mg)
- Paracetamol (Active Comparator): (500 mg, 4x1)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Dexketoprofen Trometamol + Thiocolchicoside — Dexketoprofen Trometamol + Thiocolchicoside (25mg + 4mg) is a NSAID. It was given to the patients twice a day.
  Arms: Dexketoprofen Trometamol + Thiocolchicoside
Drug: Dexketoprofen Trometamol + Paracetamol — Dexketoprofen Trometamol + Paracetamol (25mg + 300mg) is a NSAID. It was given to the patients twice a day.
  Arms: Dexketoprofen Trometamol + Paracetamol
Drug: Dexketoprofen Trometamol (25mg) — Dexketoprofen Trometamol (25mg) is a NSAID. It was given to the patients twice a day.
  Arms: Dexketoprofen Trometamol
Drug: Paracetamol — Paracetamol (500 mg) is a mild analgesic and antipyretic. It was given to the patients to take only if needed as max. dose 2000mg.
  Arms: Paracetamol

SUMMARY:
The most important step in the treatment of TMJ (temporomandibular joint) disease in clinical dentistry is diagnosis and planning. The clinical findings, drug requirement and biological risk of the patients determine the examination methods to be used in the Treatment of Temporomandibular Joint Disorders. In this context, it is thought that studies in the field of dentistry should be increased in order to increase the success in the treatment of TMJ Disorders. The aim of the study is to evaluate the efficacy of of different pain relievers as Dexketoprofen Trometamol + Thiocolchicoside, dexketoprofen trometamol + paracetamol and Dexketoprofen Trometamol in the treatment of pain in TMJ disorders.

DETAILED DESCRIPTION:
The study was carried out on 200 patients aged 18 and over, who applied to Van Yuzuncu Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, with complaints of pain due to temporomandibular disease. When patients first applied to the clinic, their anamnesis were taken and they were directed to MR (Magnetic Resonance) imaging after clinical evaluation. Patients who meet the inclusion criteria and volunteer were included in the study. Patients were randomly divided into 4 groups. Medications were given to patients by auxiliary staff and the study was double-blind. Medicines were given as follows. Dexketoprofen Trometamol + Thiocolchicoside (25mg + 4mg, 2x1) in the 1st group, Dexketoprofen Trometamol + Paracetamol (25mg + 300mg, 2x1) in the 2nd group, only Dexketoprofen Trometamol (25mg, 2x1) in the 3rd group and paracetamol 500 mg in the 4th control group (4x1) were given. In addition, patients in each group used occlusal plate for a minimum of 8 hours per day (at night). Medicines were used regularly for 2 weeks. Paracetamol 500 mg was used only if needed for the next 2 weeks. The pain values of the patients was evaluated with the VAS scale, and the amount of mouth opening was evaluated by measuring the distance between the incisal edges of the lower and upper central teeth. Evaluations have been done at the beginning of the treatment and at the 1st week, 2nd week, 1st month and the 3rd month and the findings were recorded. After the 1st month, the patients were followed up to the 3rd month and the treatment of those who need additional treatment were continued. Obtained data will be analyzed and evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 and over
2. Individuals without any systemic disease
3. Individuals without missing teeth
4. Individuals who have not used any medication in the last week
5. Individuals with normal TMJ MR imaging
6. Patients who applied to our clinic and had pain due to temporomandibular disease.

Exclusion Criteria:

1. Individuals who do not come to their check-ups regularly
2. Individuals allergic to any of the study drugs
3. Pregnant and lactating individuals

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | 1st week
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 2nd week
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 1st month
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 3rd month
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Trismus Evaluation | 1st week
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | 2nd week
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | 1st month
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | 3rd month
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Pain Evaluation (at masticatory muscles by palpation) | 1st week
  The presence of pain in the masticatory muscles was evaluated by palpation of the muscles.
Pain Evaluation (at masticatory muscles by palpation) | 2nd week
  The presence of pain in the masticatory muscles was evaluated by palpation of the muscles.
Pain Evaluation (at masticatory muscles by palpation) | 1st month
  The presence of pain in the masticatory muscles was evaluated by palpation of the muscles.
Pain Evaluation (at masticatory muscles by palpation) | 3rd month
  The presence of pain in the masticatory muscles was evaluated by palpation of the muscles.
Clicking-Crepitus Evaluation | 1st week
  Presence or absence of clicking and/or crepitus sounds detected with auscultation at temporomandibular joint.
Clicking-Crepitus Evaluation | 2nd week
  Presence or absence of clicking and/or crepitus sounds detected with auscultation at temporomandibular joint.
Clicking-Crepitus Evaluation | 1st month
  Presence or absence of clicking and/or crepitus sounds detected with auscultation at temporomandibular joint.
Clicking-Crepitus Evaluation | 3rd month
  Presence or absence of clicking and/or crepitus sounds detected with auscultation at temporomandibular joint.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ciğerim, Assoc.Prof., Study Director — Van Yuzuncu Yil University, Faculty of Dentistry
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05529290/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05529290/ICF_001.pdf